CLINICAL TRIAL: NCT06111885
Title: Randomized, Double-blind, Crossover Trial Assessing the Efficacy of Indapamide and Chlorthalidone Compared to Hydrochlorothiazide for the Reduction of Urine Supersaturation for Kidney Stone Prevention
Brief Title: Indapamide and Chlorthalidone to Reduce Urine Supersaturation for Kidney Stone Prevention
Acronym: INDAPACHLOR
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: Department of clinical research, Bern (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: INDAPACHLOR Trial
Record Dates: First submitted 2023-10-26; First posted 2023-11-01 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Kidney Stone
Keywords: Nephrolithiasis; Kidney stones; Thiazide; Hydrochlorothiazide; Indapamide; Chlorthalidone
MeSH Terms: conditions — Kidney Calculi; Nephrolithiasis | interventions — Indapamide; Hydrochlorothiazide; Chlorthalidone

STUDY DESIGN:
Intervention Model Description: Eligible individuals will be randomly allocated to one of six treatment sequences with indapamide 2.5 mg, chlorthalidone 25 mg or hydrochlorothiazide 50 mg once daily per os in the morning. Active treatment phases will be 28 days each, separated by wash out periods of 28 days. Active treatment periods can be extended by a maximum of one week, wash out periods can be extended to a maximum of eight weeks.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Indapamide, hydrochlorothiazide and chlorthalidone will be provided in identically looking bottles containing identically looking capsules. All trial personnel that is involved in recruitment and care of patients, trial assessment, monitoring and statistical analyses will be blinded to the assigned trial arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- Indapamide + Hydrochlorothiazide + Chlorthalidone (Active Comparator): 1 capsule containing 2.5 mg indapamide per day for 28 days, followed by a 28 days wash out phase, followed by a second treatment phase with 1 capsule containing 50 mg hydrochlorothiazide per day for 28 days, followed by a 28 days wash out phase, followed by a third treatment phase with 1 capsule containing 25 mg chlorthalidone per day for 28 days.
  Interventions: Drug: Indapamide 2.5 MG; Drug: Hydrochlorothiazide 50Mg; Drug: Chlorthalidone 25mg
- Hydrochlorothiazide + Chlorthalidone + Indapamide (Active Comparator): 1 capsule containing 50 mg hydrochlorothiazide per day for 28 days, followed by a 28 days wash out phase, followed by a second treatment phase with 1 capsule containing 25 mg chlorthalidone per day for 28 days, followed by a 28 days wash out phase, followed by a third treatment phase with 1 capsule containing 2.5 mg indapamide per day for 28 days.
  Interventions: Drug: Indapamide 2.5 MG; Drug: Hydrochlorothiazide 50Mg; Drug: Chlorthalidone 25mg
- Chlorthalidone + Indapamide + Hydrochlorothiazide (Active Comparator): 1 capsule containing 25 mg chlorthalidone per day for 28 days, followed by a 28 days wash out phase, followed by a second treatment phase with 1 capsule containing 2.5 mg indapamide per day for 28 days, followed by a 28 days wash out phase, followed by a third treatment phase with 1 capsule containing 50 mg hydrochlorothiazide per day for 28 days.
  Interventions: Drug: Indapamide 2.5 MG; Drug: Hydrochlorothiazide 50Mg; Drug: Chlorthalidone 25mg
- Hydrochlorothiazide + Indapamide + Chlorthalidone (Active Comparator): 1 capsule containing 50 mg hydrochlorothiazide per day for 28 days, followed by a 28 days wash out phase, followed by a second treatment phase with 1 capsule containing 2.5 mg indapamide per day for 28 days, followed by a 28 days wash out phase, followed by a third treatment phase with 1 capsule containing 25 mg chlorthalidone per day for 28 days.
  Interventions: Drug: Indapamide 2.5 MG; Drug: Hydrochlorothiazide 50Mg; Drug: Chlorthalidone 25mg
- Indapamide + Chlorthalidone + Hydrochlorothiazide (Active Comparator): 1 capsule containing 2.5 mg indapamide per day for 28 days, followed by a 28 days wash out phase, followed by a second treatment phase with 1 capsule containing 25 mg chlorthalidone per day for 28 days, followed by a 28 days wash out phase, followed by a third treatment phase with 1 capsule containing 50 mg hydrochlorothiazide per day for 28 days.
  Interventions: Drug: Indapamide 2.5 MG; Drug: Hydrochlorothiazide 50Mg; Drug: Chlorthalidone 25mg
- Chlorthalidone + Hydrochlorothiazide + Indapamide (Active Comparator): 1 capsule containing 25 mg chlorthalidone per day for 28 days, followed by a 28 days wash out phase, followed by a second treatment phase with 1 capsule containing 50 mg hydrochlorothiazide per day for 28 days, followed by a 28 days wash out phase, followed by a third treatment phase with 1 capsule containing 2.5 mg indapamide per day for 28 days.
  Interventions: Drug: Indapamide 2.5 MG; Drug: Hydrochlorothiazide 50Mg; Drug: Chlorthalidone 25mg

INTERVENTIONS:
Drug: Indapamide 2.5 MG — 1 indapamide 2.5 mg capsule per day for 28 days
Drug: Hydrochlorothiazide 50Mg — 1 hydrochlorothiazide 50 mg capsule per day for 28 days
Drug: Chlorthalidone 25mg — 1 chlorthalidone 25 mg capsule per day for 28 days

SUMMARY:
The aim of this study is to test the efficacy of the two long-acting thiazide-like diuretics indapamide and chlorthalidone in reducing urine supersaturation for calcium oxalate and calcium phosphate compared to the short-acting thiazide diuretic hydrochlorothiazide for the prevention of calcium-containing kidney stones.

DETAILED DESCRIPTION:
Background and Rationale:

Kidney stones are the most common condition affecting the kidney. Both prevalence and incidence are increasing rapidly, driven by global warming, urbanization, dietary habits and occupational changes. Kidney stones are highly recurrent, associated with increased mortality, significant morbidity and reduced quality of life, and result in enormous health care expenditures. Hence, effective preventive measures are an undisputed medical need. Thiazide and thiazide-like diuretics ("thiazides") have been the cornerstone of pharmacologic recurrence prevention since >50 years. The NOSTONE trial (NCT03057431), the only state-of-the-art trial ever performed for pharmacologic recurrence prevention, recently revealed that the most widely prescribed and best studied thiazide, hydrochlorothiazide, is not effectively preventing kidney stone recurrence. If these results also apply to the two more potent and long-acting thiazide-like diuretics indapamide and chlorthalidone is currently unknown. No head-to-head comparison of different thiazides for prevention of kidney stone recurrence has ever been performed. Thus, the role of thiazides in the prevention of kidney stone recurrence remains unclear. This poses the urgent need for a clinical trial that addresses this critical knowledge gap.

Objective:

The investigators plan to conduct a single-center, prospective, randomized, double-blind, crossover trial (INDAPACHLOR) to assess if indapamide and chlorthalidone are superior to hydrochlorothiazide in reducing urine supersaturations of calcium oxalate and calcium phosphate, the two best validated biochemical indicators of kidney stone recurrence risk.

Methodology:

Patients will be allocated to indapamide 2.5 mg once daily, chlorthalidone 25 mg once daily and hydrochlorothiazide 50 mg once daily in a random sequence. The three consecutive active treatment periods of 4 weeks each will be separated by wash-out periods of 4 weeks. The investigators will include 99 adult (>18 years old) patients with recurrent (≥ 2 stone episodes in the last 10 years) calcium-containing kidney stones (containing ≥ 50% of calcium oxalate, calcium phosphate or a mixture of both). All patients will receive a state-of-the art concomitant non-pharmacologic intervention to prevent stone recurrence according to current guidelines. The primary outcome will be reduction of urine supersaturations of calcium oxalate and calcium phosphate at 4 weeks with indapamide or chlorthalidone compared to hydrochlorothiazide. Secondary outcomes will be changes in 24-hour urine and blood parameters, ambulatory blood pressure and adverse events elicited by indapamide or chlorthalidone compared to hydrochlorothiazide. In an exploratory outcome, the abundance of the thiazide target, the sodium/chloride co-transporter, will be analyzed in urinary extracellular vesicles at 4 weeks.

Expected significance:

INDAPACHLOR will provide long-sought evidence on the comparative efficacy of commonly used thiazides in lowering urine supersaturations and is thus expected to have a strong guideline-changing impact, which will transform patient care for this very common disease.

ELIGIBILITY:
Inclusion criteria:

* Written, informed consent.
* Age 18 years or older.
* Recurrent kidney stone disease (≥2 kidney stone episodes in the last 10 years prior to randomisation).
* Past kidney stone containing ≥50 % CaOx, CaP, or a mixture of both.

Exclusion criteria:

* Patients with secondary causes of recurrent calcium kidney stones including severe eating disorders (anorexia or bulimia), chronic bowel disease, intestinal or bariatric surgery, sarcoidosis, primary hyperparathyroidism, chronic urinary tract infection.
* Patients with the following medications: Thiazide or loop diuretics, carbonic anhydrase inhibitors (including topiramate), xanthine oxidase inhibitors, alkali, active vitamin D (calcitriol or similar), calcium supplementation, bisphosphonates, denusomab, teriparatide, sodium-glucose co-transporter 2 (SGLT2) inhibitors, strong CYP3A4 inhibitors or inducers (may affect indapamide metabolism), lithium (To be eligible for study participation, patients taking any of the above listed medications at screening must be willing to discontinue these medications at least 28 days before randomization).
* Patients with chronic kidney disease (defined as CKD-EPI eGFR <30 mL/min).
* Patients with glomerulonephritis.
* Patients with the following biochemical imbalances: severe hypercalcemia (>2.8 mmol/L), therapy-resistant hypokalemia or conditions with increased potassium loss, severe hyponatremia (<130 mmol/L), symptomatic hyperuricemia.
* Patients with hepatic encephalopathy or severe liver insufficiency.
* Patients with severe cardiac insufficiency.
* Patient with a recent cerebrovascular event.
* Patients with a solid organ transplant.
* Pregnant and lactating women (A urine pregnancy test must be performed for women of child-bearing potential, defined as women who are not surgically sterilized/hysterectomized, and/or who are postmenopausal for less than 12 months).
* Previous (within 3 months prior to randomization) or concomitant participation in another interventional clinical trial.
* Previous participation in INDAPACHLOR.
* Inability to understand and follow the protocol.
* Allergy to any one of the study drugs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Primary outcome component 1 - calcium oxalate supersaturation in urine | Calcium oxalate supersaturation will be determined at day 28 of each active treatment phase
  The trial has two primary outcomes that will be assessed separately.
  Change from baseline urine calcium oxalate supersaturation to end of treatment.
  Calcium oxalate supersaturation will be calculated by the Equil2 program.
Primary outcome component 2 - calcium phosphate supersaturation in urine | Calcium phosphate supersaturation will be determined at day 28 of each active treatment phase
  The trial has two primary outcomes that will be assessed separately.
  Change from baseline urine calcium phosphate supersaturation to end of treatment.
  Calcium phosphate supersaturation will be calculated by the Equil2 program.

SECONDARY OUTCOMES:
Blood sodium level change from baseline | Data collected at baseline and at day 28 of each active treatment phase
  Sodium level measured in mmol/l
Blood potassium level change from baseline | Data collected at baseline and at day 28 of each active treatment phase
  Potassium level measured in mmol/l
Blood chloride level change from baseline | Data collected at baseline and at day 28 of each active treatment phase
  Chloride level measured in mmol/l
Blood calcium level change from baseline | Data collected at baseline and at day 28 of each active treatment phase
  Calcium level measured in mmol/l
Blood magnesium level change from baseline | Data collected at baseline and at day 28 of each active treatment phase
  Magnesium level measured in mmol/l
Blood phosphate level change from baseline | Data collected at baseline and at day 28 of each active treatment phase
  Phosphate level measured in mmol/l
Venous bicarbonate level change from baseline | Data collected at baseline and at day 28 of each active treatment phase
  Venous bicarbonate level measured in mmol/l
Venous pH change from baseline | Data collected at baseline and at day 28 of each active treatment phase
  Venous pH measured in pH units
Venous pCO2 change from baseline | Data collected at baseline and at day 28 of each active treatment phase
  Venous pCO2 measured in mmHg
Blood glucose level change from baseline | Data collected at baseline and at day 28 of each active treatment phase
  Glucose level measured in mmol/l
Blood creatinine level change from baseline | Data collected at baseline and at day 28 of each active treatment phase
  Creatinine level measured in μmol/l
Blood urea level change from baseline | Data collected at baseline and at day 28 of each active treatment phase
  Urea level measured in mmol/l
Blood uric acid level change from baseline | Data collected at baseline and at day 28 of each active treatment phase
  Uric acid level measured in μmol/l
Blood albumin level change from baseline | Data collected at baseline and at day 28 of each active treatment phase
  Albumin level measured in g/l
Blood total cholesterol level change from baseline | Data collected at baseline and at day 28 of each active treatment phase
  Total cholesterol level measured in mmol/l
Blood HDL cholesterol level change from baseline | Data collected at baseline and at day 28 of each active treatment phase
  HDL cholesterol level measured in mmol/l
Blood LDL cholesterol level change from baseline | Data collected at baseline and at day 28 of each active treatment phase
  LDL cholesterol level measured in mmol/l
Blood triglyceride level change from baseline | Data collected at baseline and at day 28 of each active treatment phase
  Triglycerides level measured in mmol/l
Blood haemoglobin A1c level change from baseline | Data collected at baseline and at day 28 of each active treatment phase
  Haemoglobin A1c activity level measured in mU/l
Urine sodium excretion change from baseline | Data collected at baseline and at day 28 of each active treatment phase
  Urine sodium excretion measured in mmol/24 h
Urine potassium excretion change from baseline | Data collected at baseline and at day 28 of each active treatment phase
  Urine potassium excretion measured in mmol/24 h
Urine chloride excretion change from baseline | Data collected at baseline and at day 28 of each active treatment phase
  Urine chloride excretion measured in mmol/24 h
Urine calcium excretion change from baseline | Data collected at baseline and at day 28 of each active treatment phase
  Urine calcium excretion measured in mmol/24 h
Urine phosphate excretion change from baseline | Data collected at baseline and at day 28 of each active treatment phase
  Urine phosphate excretion measured in mmol/24 h
Urine magnesium excretion change from baseline | Data collected at baseline and at day 28 of each active treatment phase
  Urine magnesium excretion measured in mmol/24 h
Urine urea excretion change from baseline | Data collected at baseline and at day 28 of each active treatment phase
  Urine urea excretion measured in mmol/24 h
Urine creatinine excretion change from baseline | Data collected at baseline and at day 28 of each active treatment phase
  Urine creatinine excretion measured in μmol/24 h
Urine uric acid excretion change from baseline | Data collected at baseline and at day 28 of each active treatment phase
  Urine uric acid excretion measured in μmol/24 h
Urine citrate excretion change from baseline | Data collected at baseline and at day 28 of each active treatment phase
  Urine citrate excretion measured in mmol/24 h
Urine sulfate excretion change from baseline | Data collected at baseline and at day 28 of each active treatment phase
  Urine sulfate excretion measured in mmol/24 h
Urine oxalate excretion change from baseline | Data collected at baseline and at day 28 of each active treatment phase
  Urine oxalate excretion measured in μmol/24 h
Urine ammonium excretion change from baseline | Data collected at baseline and at day 28 of each active treatment phase
  Urine ammonium excretion measured in mmol/24 h
Urine bicarbonate excretion change from baseline | Data collected at baseline and at day 28 of each active treatment phase
  Urine bicarbonate excretion measured in mmol/24 h
Urine titratable acidity excretion change from baseline | Data collected at baseline and at day 28 of each active treatment phase
  Urine titratable acidity excretion measured in mEq/24 h
Urine pH change from baseline | Data collected at baseline and at day 28 of each active treatment phase
  pH measured in pH units

OTHER OUTCOMES:
Abundance of total sodium/chloride co-transporter (SLC12A3) in urinary extracellular vesicles | Data collected at baseline and at day 28 of each active treatment phase
  Abundance of total sodium/chloride co-transporter (SLC12A3) detected by immunoblotting on urinary extracellular vesicles, normalized to the abundance of the urinary extracellular vesicle protein Alix
Abundance of phosphorylated sodium/chloride co-transporter (SLC12A3) in urinary extracellular vesicles | Data collected at baseline and at day 28 of each active treatment phase
  Abundance of phosphorylated sodium/chloride co-transporter (SLC12A3) detected by immunoblotting on urinary extracellular vesicles, normalized to the abundance of the urinary extracellular vesicle protein Alix

CONTACTS AND LOCATIONS:
Overall Officials: Daniel G Fuster, M.D., Principal Investigator — Department of Nephrology and Hypertension, Inselspital, Bern University Hospital, Bern Switzerland
Locations (1):
- Inselspital, Department of Nephrology and Hypertension, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No
Once results have been published, trial data will be accessible to external researchers and coded datasets corresponding to each publication will be made available. Investigators wishing to replicate the analyses or to do an individual patient meta-analysis may request the data to the Sponsor-Investigator.

REFERENCES:
- [Derived] Scoglio M, Bargagli M, Rintelen F, Roumet M, Trelle S, Fuster DG. Indapamide or chlorthalidone to reduce urine supersaturation for secondary prevention of kidney stones: protocol for a randomised, double-blind, cross-over trial (INDAPACHLOR). BMJ Open. 2025 Jun 16;15(6):e101594. doi: 10.1136/bmjopen-2025-101594. PMID 40523783